CLINICAL TRIAL: NCT07190599
Title: Effects of Neuromuscular Electrical Stimulation Combined With Proprioceptive Neuromuscular Facilitation in Adults With a History of Ankle Sprain
Brief Title: NMES With PNF for Ankle Sprain Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fooyin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCKU HREC-E-114-0093-2
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-09

CONDITIONS: Ankle Sprain
Keywords: Ankle sprain; Balance; Proprioception; Strength; Pain; Range of motion
MeSH Terms: conditions — Ankle Injuries; Pain | interventions — Muscle Stretching Exercises; Single Person

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NMES with PNF (Experimental): The experimental group will receive proprioceptive neuromuscular facilitation (PNF) stretching combined with neuromuscular electrical stimulation (NMES)
  Interventions: Behavioral: Proprioceptive neuromuscular facilitation (PNF) with neuromuscular electrical stimulation (NMES)
- PNF only (Active Comparator): The control group will receive PNF stretching only.
  Interventions: Behavioral: Proprioceptive neuromuscular facilitation (PNF) only

INTERVENTIONS:
Behavioral: Proprioceptive neuromuscular facilitation (PNF) with neuromuscular electrical stimulation (NMES) — The NMES was applied during the plantarflexor contraction phase of the PNF stretching (described as below). Two electrodes (4 × 8 cm) were used for stimulation, placed on the triceps surae of the affected side: one positioned 5 cm below the popliteal fossa, and the other placed 5 cm below the first electrode, directly over the triceps surae. The hold-relax technique of proprioceptive neuromuscular facilitation (PNF) will be applied to stretch the triceps surae muscle. It will be performed ten times on the affected limb during each treatment session, lasting approximately 10 minutes in total. Participants will receive interventions three times per week for four weeks, for a total of twelve sessions.
  Arms: NMES with PNF
Behavioral: Proprioceptive neuromuscular facilitation (PNF) only — The hold-relax technique will be applied to stretch the triceps surae muscle. It will be performed ten times on the affected limb during each treatment session, lasting approximately 10 minutes in total. Participants will receive interventions three times per week for four weeks, for a total of twelve sessions.
  Arms: PNF only

SUMMARY:
Ankle sprains are one of the most common sports injuries. In some people, they can lead to chronic ankle problems that affect daily life and sports performance. In this study, we want to see if combining neuromuscular electrical stimulation (NMES) with proprioceptive neuromuscular facilitation (PNF) can help improve these problems. We plan to recruit 60 participants, with 30 in the experimental group and 30 in the control group. The experimental group will receive PNF stretching with NMES, while the control group will only do PNF stretching. Both groups will have training three times a week for four weeks (12 sessions in total). We will test participants before and after the program, looking at pain, balance, range of motion, proprioception, strength, joint mobility, and functional limitations. We expect that 12 sessions will help improve chronic ankle problems, and that NMES combined with PNF will be more effective than PNF alone.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-30 years
* Adults with a history of ankle sprain

Exclusion Criteria:

* Participants with ankle fractures, dislocations, grade III ankle sprains, bony restrictions, swelling, neuropathy, or any other neuromuscular disorders are excluded.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Star Excursion Balance Test, SEBT | 1. Baseline (Day 1, prior to intervention) 2. Post-intervention (after 12 sessions, Week 4)
  Balance ability will be assessed using the Star Excursion Balance Test (SEBT). Participants stand barefoot at the center of a grid with eight lines extending at 45° angles. They are instructed to reach with the distal part of the foot to touch the farthest point along each line while maintaining a standing position. The examiner recorded the reached distance in centimeters, measured from the center of the grid to the point touched by the participant's big toe.
Proprioception - ankle dorsiflexion (degrees) | 1. Baseline (Day 1, prior to intervention) 2. Post-intervention (after 12 sessions, Week 4)
  Proprioception of the affected ankle will be measured using the Micro FET3 inclinometer. The examiner moves the foot to a target angle (hold for 10 seconds), and then returned to the starting position. Participants then actively reproduces the angle. The difference between the target and reproduced angles represented proprioceptive accuracy.
Proprioception - ankle plantarflexion (degrees) | 1. Baseline (Day 1, prior to intervention) 2. Post-intervention (after 12 sessions, Week 4)
  Proprioception of the affected ankle will be measured using the Micro FET3 inclinometer. The examiner moves the foot to a target angle (hold for 10 seconds), and then returned to the starting position. Participants then actively reproduces the angle. The difference between the target and reproduced angles represented proprioceptive accuracy.
Muscle strength - ankle dorsiflexors (kg) | 1. Baseline (Day 1, prior to intervention) 2. Post-intervention (after 12 sessions, Week 4)
  A dynamometer (Micro FET3) will be placed on the dorsal surfaces of the metatarsals to measure strength of dorsiflexors.
Muscle strength - ankle plantarflexors (kg) | 1. Baseline (Day 1, prior to intervention) 2. Post-intervention (after 12 sessions, Week 4)
  A dynamometer (Micro FET3) will be placed on the plantar surfaces of the metatarsals to measure strength of plantarflexors.
Range of motion - Ankle dorsiflexion (degrees) | 1. Baseline (Day 1, prior to intervention) 2. Post-intervention (after 12 sessions, Week 4)
  The axis of the goniometer was placed at the lateral malleolus, the stationary arm aligned with the lateral fibula, and the moving arm aligned with the fifth metatarsal. Participants will be instructed to actively move the ankle from 0° starting position to maximal dorsiflexion.
Range of motion - Ankle plantarflexion (degrees) | 1. Baseline (Day 1, prior to intervention) 2. Post-intervention (after 12 sessions, Week 4)
  The axis of the goniometer was placed at the lateral malleolus, the stationary arm aligned with the lateral fibula, and the moving arm aligned with the fifth metatarsal. Participants will be instructed to actively move the ankle from 0° starting position to maximal plantarflexion

SECONDARY OUTCOMES:
The Foot and Ankle Disability Index (FADI) | 1. Baseline (Day 1, prior to intervention) 2. Post-intervention (after 12 sessions, Week 4)
  Functional limitations will be assessed using the Foot and Ankle Disability Index (FADI). The FADI includes 22 questions related to functional activities and 4 questions related to pain. Each item is scored from 0 (unable to do) to 4 (no difficulty), with a maximum total score of 104, which is then converted to a percentage. A score of 100% indicates no functional limitation.
Knee to wall test | 1. Baseline (Day 1, prior to intervention) 2. Post-intervention (after 12 sessions, Week 4)
  Participants stand facing a wall with their toes about 10 cm away. The non-affected foot steps back, and the affected knee bends forward to touch the wall while keeping the heel on the ground. If the knee cannot reach the wall, the front foot moves closer. The distance from the affected big toe to the wall is then measured. The distance (cm) from the participant's big toe of the affected foot to the wall was measured and recorded.
Visual analog scale (VAS) | 1. Baseline (Day 1, prior to intervention) 2. Post-intervention (after 12 sessions, Week 4)
  Participants mark their pain level on a 10-cm line, with the left end representing 'no pain' and the right end representing 'unbearable pain.' The mark indicates the intensity of their pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Fooyin University, Kaohsiung City, No. 151, Jinxue Road, Daliao District, Taiwan

IPD SHARING:
Plan to Share IPD: No